CLINICAL TRIAL: NCT03608228
Title: Invasive Approach to Model Human Cortex-Basal Ganglia Action-Regulating Networks
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: The Cleveland Clinic (Other); University of California, San Francisco (Other); University of California, San Diego (Other); California Institute of Technology (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-001516
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease Patients Undergoing Deep Brain Stimulation (DBS) Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease
  Interventions: Other: Measuring electrical signals from the brain

INTERVENTIONS:
Other: Measuring electrical signals from the brain — If patients participate in this study, after the deep brain stimulator leads have been implanted, the researcher(s) will plan to measure electrical signals from the brain while patients perform hand movement tasks.

SUMMARY:
The brain networks controlling movement are complex, involving multiple areas of the brain. Some neurological diseases, like Parkinson's disease, cause abnormalities in the brain networks. Deep brain stimulation is a treatment that is used to treat these types of neurological diseases. Through this research, the investigators will take advantage of the unique opportunity provided by awake deep brain stimulation surgery to learn more about how the brain functions in a diseased state and how deep brain stimulation changes these networks. This study aims to enroll up to 75 subjects over a period of 2.5 years. Those who participate in the study will spend up to 40 minutes during their deep brain stimulation surgery during which researchers will record signals from deep structures within the brain as well as the surface of the brain using electrodes that are temporarily placed for research purposes. During the study, researchers will record signals while subjects perform three different tasks, in some cases while the brain is stimulated. Study participation is limited to the intraoperative environment with no additional study visits required.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Rigid-akinetic subtype of Parkinson's disease, diagnosed by a movement disorders neurologist
3. Clinical indications, as deemed by a multidisciplinary team of neurologists and neurosurgeons, for deep brain stimulation surgery, including motor fluctuations, difficult-to-control-dyskinesias, unpredictable off-times, and/or dystonia
4. Preoperative MRI without cortical or subdural adhesions or vascular abnormalities
5. Subject is medically fit for surgical intervention, as deemed by a primary care physician

Exclusion Criteria:

1. Inability or unwillingness to tolerate 20 minutes and up to 40 minutes of additional operative time
2. Patient with history of secondary Parkinsonism, stroke, or progressive central nervous system disease other than Parkinson's disease.
3. Subject is at high risk for surgical complications such as active systemic infection, coagulation disorders (such as the use of anti-thrombotic therapies) or platelet count below 100,000.
4. Subject is taking chronic anticoagulants or antiplatelet agent or subject has an abnormally elevated preoperative coagulation profile (either (Partial Thromboplastin Time) PTT or prothrombin time/INR).
5. Patients with recent use (within one week) of anticoagulant or antiplatelet agent use
6. Subject has history of bleeding or immune compromise.
7. Subject has history of implant-related infection.
8. Subject has a prior history of seizures or epilepsy.
9. Subject has a clinically significant or unstable medical condition including uncontrolled systemic hypertension with values above 170/100; cardiac or pulmonary disease; uncorrected coagulation abnormalities; diabetes; or any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.
10. Subject has a significant abnormality on preoperative brain MRI
11. Subject has had prior craniotomy or brain surgery.
12. Subject has significant memory impairment (based on Montreal Cognitive Assessment (MoCA) < 23).
13. Subject has a disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

    1. Cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease
    2. Does not speak a principal language associated with the region
    3. Hearing loss that prevents adequate communication with researchers.
14. Subject has moderate or severe depression (HAMD ≥ 17)
15. Subject is implanted with any neuromodulation device in the head including, but not limited to cochlear implant, deep brain stimulator, or auditory brain implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are patients who are undergoing deep brain stimulation implantation for treatment of Parkinson's disease based on clinical indications as determined by a multidisciplinary neurology-neurosurgery team at each center.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Differences in neural signals related to stopping and conflicting movements | Up to 40 minutes
  Patients will be asked to perform hand movements in response to either a go signals, a conflict signal, or a stopping signal.

CONTACTS AND LOCATIONS:
Locations (1):
- Nader Pouratian, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No